CLINICAL TRIAL: NCT06859463
Title: Muscle Function and Tenderness in Migraine, Tension-Type Headache, and Posttraumatic Headache Patients: a Cross-Sectional Study
Brief Title: Muscle Function and Tenderness Differences in Headache Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Bjarne Kjeldgaard Madsen, physiotherapist ph.d, Danish Headache Center
Other Study IDs: F-24075902
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Migraine; Tension Headache; Posttraumatic Headache
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache; Post-Traumatic Headache

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Migraine patients Migraine patients with at least 10 days per month of headache: Tensional-type headache patients Tensional-type headache patients with at least 10 days per month of headache.
  Interventions: Device: Muscle function
- Posttraumatic headache patients Posttraumatic headache patients with at least 10 days per month of h
  Interventions: Device: Muscle function
- Tensional-type headache patients Tensional-type headache patients with at least 10 days per month of
  Interventions: Device: Muscle function

INTERVENTIONS:
Device: Muscle function — Functional evaluation First, the patients will fill the Fysisk Aktivitet Questionnaire, the o Klinisk Oral Fysiologi (KU) Questionnaire and the Harvard Trauma Questionnaire. Then, the evaluator will applicate the Total Tenderness Score (TTS) for evaluating their tenderness in different spots of the head and neck regions. The next evaluation comprehends the evaluation of the maximal voluntary isometric contraction (MVIC) for the different neck movements and the rate of force development (RFD) of the shoulder elevation. After this, patients will perform the cranio-cervical flexion test (CCFT), and, finally, the Ito test to evaluate the lumbar endurance.

SUMMARY:
This cross-sectional study aims to compare muscle function of the neck, and shoulder and muscle tenderness in three groups of headache patients: migraine, tension-type headache, and posttraumatic headache. The study will evaluate muscle tenderness through the Total Tenderness Score (TTS) and muscle function through maximum voluntary isometric contraction (MVIC) and rate of force development (RFD). Additionally, functional assessments such as the Cranio-Cervical Flexion Test (CCFT) and Ito Test will be performed.

ELIGIBILITY:
Inclusion Criteria:Criteria: Inclusion Criteria:

* Aged 18 to 65 years.
* Diagnosis of migraine, tension-type headache, or posttraumatic headache, occurring at least 10 days per month.
* For tension-type headache patients, maximum of 3 days per month with migraine.

Exclusion Criteria:

* Pregnancy.
* Significant psychiatric comorbidities (e.g., severe depression).
* Medication-overuse headache.
* Severe osteoarthritis in the neck or shoulder, or cervical disc herniation.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Migraine, tensional-type headache, and posttraumatic headache patients who are between 18-65 years old and have at least 10 days of headache per month
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure: 1.Rate of Force Development (RFD) | 1 year
  Rate of Force Development (RFD) of the shoulder elevation Maximum voluntary isometric contraction performed "as fast and hard as possible" using a custom dynamometer for the shoulder elevation movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Copenhagen, Region H, Denmark